CLINICAL TRIAL: NCT04558034
Title: The Use of Cryotherapy to Prevent Paclitaxel-induced Peripheral Neuropathy and Nail Changes in Women With Breast Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator retired before study completed.
Sponsor: Parkview Health (Other)
Responsible Party: Principal Investigator, Danielle Payne, Prinicipal Investigator, Parkview Health
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NUR20-0124CRYO
Record Dates: First submitted 2020-09-03; First posted 2020-09-22 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Cryotherapy Effect; Peripheral Neuropathy; Nail Toxicity
MeSH Terms: conditions — Peripheral Nervous System Diseases | interventions — Cryotherapy

STUDY DESIGN:
Intervention Model Description: There are 2 arms to the study.The Elasto-gel mitt and Rapid Relief slipper will be placed either on one hand/foot or both based on the patient's medical oncologist. All subjects will have a standardized onset/duration of therapy which includes the following :
  * 15 minutes prior to the paclitaxel infusion,
  * Continuously during the paclitaxel infusion,
  * 15 minutes after completion of paclitaxel for a total of 90 minutes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventioncryotherapy/control (Active Comparator): Subjects will have one mitt/one slipper and serve as their own control
  Interventions: Other: cryotherapy
- standard of care (No Intervention): Subjects will have two mitts/slippers

INTERVENTIONS:
Other: cryotherapy — cryotherapy will be delivered
  Arms: Interventioncryotherapy/control

SUMMARY:
This study will determine the efficacy of cryotherapy to prevent paclitaxel-induced peripheral neuropathy and nail changes in women with breast cancer.

DETAILED DESCRIPTION:
Women with breast cancer receiving paclitaxel will complete the Brief Pain Inventory(BPI), Neuropathic Pain Syndrome Inventory (NPSI)while a member of the research team will conduct an assessment of their nails. Once complete, cryotherapy will be administered 15 minutes prior to the paclitaxel infusion, continuously during and then 15 minutes after completion of the paclitaxel for a total of 90 minutes. Cyrotherapy will be delivered using Elasto-gel mitts and Rapid relief slippers. These items will be changed 45min after initiation to ensure coldness.

There will be two arms of the study. One arm will include subjects who will wear one slipper/one mitt on their foot/hand while the other foot/hand will serve as a control. The other arm will include subjects who will have cryotherapy to both hands and feet. . This process will be repeated for a total of 12 times in conjunction with 12 doses of paclitaxel. At time point 13, during a routine visit to their oncologist, the subjects nails will be reassessed along with completion of the BPI and NPSIA total of 25 subjects will be enrolled in each arm.

ELIGIBILITY:
Inclusion Criteria:

* Females 18 or older
* Histologically confirmed diagnosis of breast cancer
* Receiving neo-adjuvant or adjuvant dose-dense anthracycline (AC) plus taxane-based chemotherapy or paclitaxel in combination with trastuzumab and pertuzumab

Exclusion Criteria:

* Prior taxane therapy
* Prior oxaliplatin therapy
* Non-English speaking
* History of peripheral neuropathy, i.e., Buerger's disease
* History of diabetes mellitus
* Pre-existing peripheral neuropathy from other conditions, e.g., Raynaud's disease, Guillain-Barre, Miller Fisher Syndrome
* Hand, nail or foot conditions, e.g., hand/foot syndrome, arthritis, hammer toe, carpal tunnel, bunions, deformities
* Alcohol abuse (history/current)
* Current medication usage of opioids, anti-depressants, anti-convulsants, glutamines, vitamin B12

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Enrollment: 14 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2021-02-03 (Actual); Study Completion 2021-02-03 (Actual)

PRIMARY OUTCOMES:
Numbness,tingling,pain ,nail toxicities | 13 weeks
  absence of numbness and tingling in the treated hands/feet
  * If there is an absence of pain in the treated hands/feet
  * If there is an absence of nail changes in the treated hands/feet

CONTACTS AND LOCATIONS:
Overall Officials: Danielle R Payne, MSN, Principal Investigator — Parkview Health
Locations (1):
- Parkview Cancer Institute, Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
The following will be shared: Individual participant data that underlie the results reported in the planned article after deidentification including text,tables,figures, appendices
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication and no end date
Access Criteria: Data will be available to anyone who wishes to access the data for any purpose by contacting nancy.ehmke@parkview.com

REFERENCES:
- [Background] Alessandrini A, Starace M, Cere G, Brandi N, Piraccini BM. Management and Outcome of Taxane-Induced Nail Side Effects: Experience of 79 Patients from a Single Centre. Skin Appendage Disord. 2019 Aug;5(5):276-282. doi: 10.1159/000497824. Epub 2019 Mar 22. PMID 31559250
- [Background] Autissier E. Chemotherapy-Induced Peripheral Neuropathy: Association With Increased Risk of Falls and Injuries. Clin J Oncol Nurs. 2019 Aug 1;23(4):405-410. doi: 10.1188/19.CJON.405-410. PMID 31322611
- [Background] Argyriou AA, Kyritsis AP, Makatsoris T, Kalofonos HP. Chemotherapy-induced peripheral neuropathy in adults: a comprehensive update of the literature. Cancer Manag Res. 2014 Mar 19;6:135-47. doi: 10.2147/CMAR.S44261. eCollection 2014. PMID 24672257
- [Background] Bandos H, Melnikow J, Rivera DR, Swain SM, Sturtz K, Fehrenbacher L, Wade JL 3rd, Brufsky AM, Julian TB, Margolese RG, McCarron EC, Ganz PA. Long-term Peripheral Neuropathy in Breast Cancer Patients Treated With Adjuvant Chemotherapy: NRG Oncology/NSABP B-30. J Natl Cancer Inst. 2018 Feb 1;110(2):djx162. doi: 10.1093/jnci/djx162. PMID 28954297
- [Background] Bouhassira D, Attal N, Fermanian J, Alchaar H, Gautron M, Masquelier E, Rostaing S, Lanteri-Minet M, Collin E, Grisart J, Boureau F. Development and validation of the Neuropathic Pain Symptom Inventory. Pain. 2004 Apr;108(3):248-257. doi: 10.1016/j.pain.2003.12.024. PMID 15030944
- [Background] Bhatnagar B, Gilmore S, Goloubeva O, Pelser C, Medeiros M, Chumsri S, Tkaczuk K, Edelman M, Bao T. Chemotherapy dose reduction due to chemotherapy induced peripheral neuropathy in breast cancer patients receiving chemotherapy in the neoadjuvant or adjuvant settings: a single-center experience. Springerplus. 2014 Jul 16;3:366. doi: 10.1186/2193-1801-3-366. eCollection 2014. PMID 25089251
- [Background] Can G, Aydiner A, Cavdar I. Taxane-induced nail changes: Predictors and efficacy of the use of frozen gloves and socks in the prevention of nail toxicity. Eur J Oncol Nurs. 2012 Jul;16(3):270-5. doi: 10.1016/j.ejon.2011.06.007. Epub 2011 Jul 23. PMID 21784705
- [Background] Capriotti K, Capriotti JA, Lessin S, Wu S, Goldfarb S, Belum VR, Lacouture ME. The risk of nail changes with taxane chemotherapy: a systematic review of the literature and meta-analysis. Br J Dermatol. 2015 Sep;173(3):842-5. doi: 10.1111/bjd.13743. Epub 2015 Jul 29. No abstract available. PMID 25704465
- [Background] Chan YN, Jheng YW, Wang PJ, Chen CY, Lin MW, Wang YJ. Taxane-Induced Peripheral Neuropathy: Objective and Subjective Comparison Between Paclitaxel and Docetaxel in Patients With Breast Cancer. Clin J Oncol Nurs. 2019 Oct 1;23(5):494-501. doi: 10.1188/19.CJON.494-501. PMID 31538967
- [Background] Cassidy J, Misset JL. Oxaliplatin-related side effects: characteristics and management. Semin Oncol. 2002 Oct;29(5 Suppl 15):11-20. doi: 10.1053/sonc.2002.35524. PMID 12422304
- [Background] Childress J, Lokich J. Cutaneous hand and foot toxicity associated with cancer chemotherapy. Am J Clin Oncol. 2003 Oct;26(5):435-6. doi: 10.1097/01.coc.0000026486.56886.18. No abstract available. PMID 14528066
- [Background] Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Ann Acad Med Singap. 1994 Mar;23(2):129-38. PMID 8080219
- [Background] Cioroiu C, Weimer LH. Update on Chemotherapy-Induced Peripheral Neuropathy. Curr Neurol Neurosci Rep. 2017 Jun;17(6):47. doi: 10.1007/s11910-017-0757-7. PMID 28421360
- [Background] Cunningham D, Gilchrist NL, Forrest GJ, Soukop M. Onycholysis associated with cytotoxic drugs. Br Med J (Clin Res Ed). 1985 Mar 2;290(6469):675-6. doi: 10.1136/bmj.290.6469.675-a. No abstract available. PMID 2578850
- [Background] Daut RL, Cleeland CS. The prevalence and severity of pain in cancer. Cancer. 1982 Nov 1;50(9):1913-8. doi: 10.1002/1097-0142(19821101)50:93.0.co;2-r. PMID 7116316
- [Background] De Giorgi U, Rosti G, Monti M, Frassineti GL, Marangolo M. Onycholysis secondary to multiple paclitaxel 1-hour infusions: possible role for its vehicle (Cremophor EL). Ann Oncol. 2003 Oct;14(10):1588-9. doi: 10.1093/annonc/mdg419. No abstract available. PMID 14504063
- [Background] Descoeur J, Pereira V, Pizzoccaro A, Francois A, Ling B, Maffre V, Couette B, Busserolles J, Courteix C, Noel J, Lazdunski M, Eschalier A, Authier N, Bourinet E. Oxaliplatin-induced cold hypersensitivity is due to remodelling of ion channel expression in nociceptors. EMBO Mol Med. 2011 May;3(5):266-78. doi: 10.1002/emmm.201100134. Epub 2011 Mar 24. PMID 21438154
- [Background] Eckhoff L, Knoop AS, Jensen MB, Ejlertsen B, Ewertz M. Risk of docetaxel-induced peripheral neuropathy among 1,725 Danish patients with early stage breast cancer. Breast Cancer Res Treat. 2013 Nov;142(1):109-18. doi: 10.1007/s10549-013-2728-2. Epub 2013 Oct 17. PMID 24132874
- [Background] Elasto-Gel(2019).Elasto-Gel.Retrieved on December 1,2019 from https://www.elastogels.com/product/elasto-gel-hot-cold-therapy-mitten/
- [Background] Forsyth PA, Balmaceda C, Peterson K, Seidman AD, Brasher P, DeAngelis LM. Prospective study of paclitaxel-induced peripheral neuropathy with quantitative sensory testing. J Neurooncol. 1997 Oct;35(1):47-53. doi: 10.1023/a:1005805907311. PMID 9266440
- [Background] Flory SM, Solimando DA Jr, Webster GF, Dunton CJ, Neufeld JM, Haffey MB. Onycholysis associated with weekly administration of paclitaxel. Ann Pharmacother. 1999 May;33(5):584-6. doi: 10.1345/aph.18307. PMID 10369623
- [Background] Gilbar P, Hain A, Peereboom VM. Nail toxicity induced by cancer chemotherapy. J Oncol Pharm Pract. 2009 Sep;15(3):143-55. doi: 10.1177/1078155208100450. Epub 2009 Jan 26. PMID 19171552
- [Background] Griffiths C, Kwon N, Beaumont JL, Paice JA. Cold therapy to prevent paclitaxel-induced peripheral neuropathy. Support Care Cancer. 2018 Oct;26(10):3461-3469. doi: 10.1007/s00520-018-4199-9. Epub 2018 Apr 21. PMID 29681015
- [Background] Grisold W, Cavaletti G, Windebank AJ. Peripheral neuropathies from chemotherapeutics and targeted agents: diagnosis, treatment, and prevention. Neuro Oncol. 2012 Sep;14 Suppl 4(Suppl 4):iv45-54. doi: 10.1093/neuonc/nos203. PMID 23095830
- [Background] Hanai A, Ishiguro H, Sozu T, Tsuda M, Yano I, Nakagawa T, Imai S, Hamabe Y, Toi M, Arai H, Tsuboyama T. Effects of Cryotherapy on Objective and Subjective Symptoms of Paclitaxel-Induced Neuropathy: Prospective Self-Controlled Trial. J Natl Cancer Inst. 2018 Feb 1;110(2):141-148. doi: 10.1093/jnci/djx178. PMID 29924336
- [Background] Hausheer FH, Schilsky RL, Bain S, Berghorn EJ, Lieberman F. Diagnosis, management, and evaluation of chemotherapy-induced peripheral neuropathy. Semin Oncol. 2006 Feb;33(1):15-49. doi: 10.1053/j.seminoncol.2005.12.010. PMID 16473643
- [Background] Hershman DL, Lacchetti C, Dworkin RH, Lavoie Smith EM, Bleeker J, Cavaletti G, Chauhan C, Gavin P, Lavino A, Lustberg MB, Paice J, Schneider B, Smith ML, Smith T, Terstriep S, Wagner-Johnston N, Bak K, Loprinzi CL; American Society of Clinical Oncology. Prevention and management of chemotherapy-induced peripheral neuropathy in survivors of adult cancers: American Society of Clinical Oncology clinical practice guideline. J Clin Oncol. 2014 Jun 20;32(18):1941-67. doi: 10.1200/JCO.2013.54.0914. Epub 2014 Apr 14. PMID 24733808
- [Background] Hoffman,K. (2014). Diagnosing and Treating Chemotherapy-Induced Nail Changes. Podiatry Today,27(2). Retrieved on December 16, 2019from https://www.podiatrytoday.com/diagnosing-and-treating-chemotherapy-induced-nail-changes
- [Background] Hussain S, Anderson DN, Salvatti ME, Adamson B, McManus M, Braverman AS. Onycholysis as a complication of systemic chemotherapy: report of five cases associated with prolonged weekly paclitaxel therapy and review of the literature. Cancer. 2000 May 15;88(10):2367-71. doi: 10.1002/(sici)1097-0142(20000515)88:103.0.co;2-#. PMID 10820360
- [Background] Ishiguro H, Takashima S, Yoshimura K, Yano I, Yamamoto T, Niimi M, Yamashiro H, Ueno T, Takeuchi M, Sugie T, Yanagihara K, Toi M, Fukushima M. Degree of freezing does not affect efficacy of frozen gloves for prevention of docetaxel-induced nail toxicity in breast cancer patients. Support Care Cancer. 2012 Sep;20(9):2017-24. doi: 10.1007/s00520-011-1308-4. Epub 2011 Nov 16. PMID 22086405
- [Background] LaPointe NE, Morfini G, Brady ST, Feinstein SC, Wilson L, Jordan MA. Effects of eribulin, vincristine, paclitaxel and ixabepilone on fast axonal transport and kinesin-1 driven microtubule gliding: implications for chemotherapy-induced peripheral neuropathy. Neurotoxicology. 2013 Jul;37:231-9. doi: 10.1016/j.neuro.2013.05.008. Epub 2013 May 24. PMID 23711742
- [Background] Lee JJ, Swain SM. Peripheral neuropathy induced by microtubule-stabilizing agents. J Clin Oncol. 2006 Apr 1;24(10):1633-42. doi: 10.1200/JCO.2005.04.0543. PMID 16575015
- [Background] Kadakia KC, Rozell SA, Butala AA, Loprinzi CL. Supportive cryotherapy: a review from head to toe. J Pain Symptom Manage. 2014 Jun;47(6):1100-15. doi: 10.1016/j.jpainsymman.2013.07.014. Epub 2013 Nov 7. PMID 24210702
- [Background] Kerckhove N, Collin A, Conde S, Chaleteix C, Pezet D, Balayssac D. Long-Term Effects, Pathophysiological Mechanisms, and Risk Factors of Chemotherapy-Induced Peripheral Neuropathies: A Comprehensive Literature Review. Front Pharmacol. 2017 Feb 24;8:86. doi: 10.3389/fphar.2017.00086. eCollection 2017. PMID 28286483
- [Background] Kolb NA, Smith AG, Singleton JR, Beck SL, Stoddard GJ, Brown S, Mooney K. The Association of Chemotherapy-Induced Peripheral Neuropathy Symptoms and the Risk of Falling. JAMA Neurol. 2016 Jul 1;73(7):860-6. doi: 10.1001/jamaneurol.2016.0383. PMID 27183099
- [Background] Kumar SP. Utilization of brief pain inventory as an assessment tool for pain in patients with cancer: a focused review. Indian J Palliat Care. 2011 May;17(2):108-15. doi: 10.4103/0973-1075.84531. PMID 21976850
- [Background] Lau CP, Hui P, Chan TC. Docetaxel-induced nail toxicity: a case of severe onycholysis and topic review. Chin Med J (Engl). 2011 Aug;124(16):2559-60. PMID 21933605
- [Background] McCarthy AL, Shaban RZ, Gillespie K, Vick J. Cryotherapy for docetaxel-induced hand and nail toxicity: randomised control trial. Support Care Cancer. 2014 May;22(5):1375-83. doi: 10.1007/s00520-013-2095-x. Epub 2013 Dec 22. PMID 24362908
- [Background] Memorial Sloan Kettering Cancer Center (2017) Nail changes during treatment with Taxane-based chemotherapy Retrieved December17,2019 from https://www.mskcc.org/pdf/cancer-care/patient-education/nail-changes-during-treatment-taxanes
- [Background] Miltenburg NC, Boogerd W. Chemotherapy-induced neuropathy: A comprehensive survey. Cancer Treat Rev. 2014 Aug;40(7):872-82. doi: 10.1016/j.ctrv.2014.04.004. Epub 2014 Apr 18. PMID 24830939
- [Background] Minisini AM, Tosti A, Sobrero AF, Mansutti M, Piraccini BM, Sacco C, Puglisi F. Taxane-induced nail changes: incidence, clinical presentation and outcome. Ann Oncol. 2003 Feb;14(2):333-7. doi: 10.1093/annonc/mdg050. PMID 12562663
- [Background] Monjazeb S, Wilson J. Epidermal Growth Factor Receptor Inhibitors: Cutaneous Side Effects and Their Management. Skin Therapy Lett. 2017 Sep;22(5):5-7. PMID 28888217
- [Background] Nicolopoulos J, Howard A. Docetaxel-induced nail dystrophy. Australas J Dermatol. 2002 Nov;43(4):293-6. doi: 10.1046/j.1440-0960.2002.00616.x. PMID 12423438
- [Background] Oncology Nursing Society.(2017). Cutaneous reactions. Retrieved on December 11, 2019 from https://www.ons.org/pep/skin-reactions
- [Background] Oncology Nursing Society.(2019). Peripheral neuropathy . Retrieved on December 11, 2019 from https://www.ons.org/pep/peripheral-neuropathy
- [Background] Park SB, Goldstein D, Krishnan AV, Lin CS, Friedlander ML, Cassidy J, Koltzenburg M, Kiernan MC. Chemotherapy-induced peripheral neurotoxicity: a critical analysis. CA Cancer J Clin. 2013 Nov-Dec;63(6):419-37. doi: 10.3322/caac.21204. PMID 24590861
- [Background] Paul LJ, Cohen PR. Paclitaxel-associated subungual pyogenic granuloma: report in a patient with breast cancer receiving paclitaxel and review of drug-induced pyogenic granulomas adjacent to and beneath the nail. J Drugs Dermatol. 2012 Feb;11(2):262-8. PMID 22270214
- [Background] Peyton L, Fischer-Cartlidge E. Extremity Cooling: A Synthesis of Cryotherapy Interventions to Reduce Peripheral Neuropathy and Nail Changes From Taxane-Based Chemotherapy. Clin J Oncol Nurs. 2019 Oct 1;23(5):522-528. doi: 10.1188/19.CJON.522-528. PMID 31538978
- [Background] Poncelet AN. An algorithm for the evaluation of peripheral neuropathy. Am Fam Physician. 1998 Feb 15;57(4):755-64. PMID 9490998
- [Background] Quasthoff S, Hartung HP. Chemotherapy-induced peripheral neuropathy. J Neurol. 2002 Jan;249(1):9-17. doi: 10.1007/pl00007853. PMID 11954874
- [Background] Rapid Aid. (2020). Cold Gel Slippers. Retrieved on March 2,2020 from http://rapidaid.com/product/hot-cold-gel-slippers/
- [Background] Robert C, Sibaud V, Mateus C, Verschoore M, Charles C, Lanoy E, Baran R. Nail toxicities induced by systemic anticancer treatments. Lancet Oncol. 2015 Apr;16(4):e181-9. doi: 10.1016/S1470-2045(14)71133-7. PMID 25846098
- [Background] Ross M, Fischer-Cartlidge E. Scalp Cooling: A Literature Review of Efficacy, Safety, and Tolerability for Chemotherapy-Induced Alopecia . Clin J Oncol Nurs. 2017 Apr 1;21(2):226-233. doi: 10.1188/17.CJON.226-233. PMID 28315539
- [Background] Sanofi (2019).Taxotere prescribing information. Retreived on December 11, 2019 from http://products.sanofi.us/taxotere/Taxotere.html
- [Background] Sato J, Mori M, Nihei S, Kumagai M, Takeuchi S, Kashiwaba M, Kudo K. The effectiveness of regional cooling for paclitaxel-induced peripheral neuropathy. J Pharm Health Care Sci. 2016 Nov 15;2:33. doi: 10.1186/s40780-016-0067-2. eCollection 2016. PMID 27891244
- [Background] Scotte F, Tourani JM, Banu E, Peyromaure M, Levy E, Marsan S, Magherini E, Fabre-Guillevin E, Andrieu JM, Oudard S. Multicenter study of a frozen glove to prevent docetaxel-induced onycholysis and cutaneous toxicity of the hand. J Clin Oncol. 2005 Jul 1;23(19):4424-9. doi: 10.1200/JCO.2005.15.651. PMID 15994152
- [Background] Scotte F, Banu E, Medioni J, Levy E, Ebenezer C, Marsan S, Banu A, Tourani JM, Andrieu JM, Oudard S. Matched case-control phase 2 study to evaluate the use of a frozen sock to prevent docetaxel-induced onycholysis and cutaneous toxicity of the foot. Cancer. 2008 Apr 1;112(7):1625-31. doi: 10.1002/cncr.23333. PMID 18286527
- [Background] Seretny M, Currie GL, Sena ES, Ramnarine S, Grant R, MacLeod MR, Colvin LA, Fallon M. Incidence, prevalence, and predictors of chemotherapy-induced peripheral neuropathy: A systematic review and meta-analysis. Pain. 2014 Dec;155(12):2461-2470. doi: 10.1016/j.pain.2014.09.020. Epub 2014 Sep 23. PMID 25261162
- [Background] Spazzapan S, Crivellari D, Lombardi D, Scuderi C, Magri MD, Veronesi A, Gatti A. Nail toxicity related to weekly taxanes: an important issue requiring a change in common toxicity criteria grading? J Clin Oncol. 2002 Nov 1;20(21):4404-5; author reply 4405. doi: 10.1200/JCO.2002.99.147. No abstract available. PMID 12409345
- [Background] Starobova H, Vetter I. Pathophysiology of Chemotherapy-Induced Peripheral Neuropathy. Front Mol Neurosci. 2017 May 31;10:174. doi: 10.3389/fnmol.2017.00174. eCollection 2017. PMID 28620280
- [Background] Sundar R, Bandla A, Tan SS, Liao LD, Kumarakulasinghe NB, Jeyasekharan AD, Ow SG, Ho J, Tan DS, Lim JS, Vijayan J, Therimadasamy AK, Hairom Z, Ang E, Ang S, Thakor NV, Lee SC, Wilder-Smith EP. Limb Hypothermia for Preventing Paclitaxel-Induced Peripheral Neuropathy in Breast Cancer Patients: A Pilot Study. Front Oncol. 2017 Jan 10;6:274. doi: 10.3389/fonc.2016.00274. eCollection 2016. PMID 28119855
- [Background] Swenson KK, Bell EM, Nissen J. Nail toxicity associated with paclitaxel treatment for ovarian cancer. Oncol Nurs Forum. 2013 Jan;40(1):17-9. doi: 10.1188/13.ONF.17-19. No abstract available. PMID 23269765
- [Background] Tofthagen C, Visovsky CM, Hopgood R. Chemotherapy-induced peripheral neuropathy: an algorithm to guide nursing management. Clin J Oncol Nurs. 2013 Apr;17(2):138-44. doi: 10.1188/13.CJON.138-144. PMID 23538249
- [Background] U.S Department of Health and Human Services (2017). Common Terminology Criteria for Adverse Events (CTCAE v. 5.0) Retrieved on December 12, 2019 from https://ctep.cancer.gov/protocoldevelopment/electronic_applications/docs/CTCAE_v5_Quick_Reference_5x7.pdf.
- [Background] Wickham R. Chemotherapy-induced peripheral neuropathy: a review and implications for oncology nursing practice. Clin J Oncol Nurs. 2007 Jun;11(3):361-76. doi: 10.1188/07.CJON.361-376. PMID 17623621
- [Background] Wildes TM, Dua P, Fowler SA, Miller JP, Carpenter CR, Avidan MS, Stark S. Systematic review of falls in older adults with cancer. J Geriatr Oncol. 2015 Jan;6(1):70-83. doi: 10.1016/j.jgo.2014.10.003. Epub 2014 Oct 30. PMID 25454770
- [Background] Wilkinson,M., Cocilovo,C., & Schar,M. (2016) Reduction of paclitaxel neuropathy with cryotherapy.Journal of Clinical Oncology.34(suppl 3S;abst 124) retrieved on December 2,2019 from https://meetinglibrary.asco.org/record/119151/abstract
- [Background] Willis, W.D (2000). The nervous system. In R.M. Berne & M.N. Levy (Eds.). Principles of physiology (pp. 68-94). St. Louis: Mosby.
- [Background] Winters-Stone KM, Horak F, Jacobs PG, Trubowitz P, Dieckmann NF, Stoyles S, Faithfull S. Falls, Functioning, and Disability Among Women With Persistent Symptoms of Chemotherapy-Induced Peripheral Neuropathy. J Clin Oncol. 2017 Aug 10;35(23):2604-2612. doi: 10.1200/JCO.2016.71.3552. Epub 2017 Jun 6. PMID 28586243